CLINICAL TRIAL: NCT04585672
Title: Ammonia Metabolism Assessed by Ammonia Infusion
Acronym: NH4 inf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-16-02-297-20
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Ammonia; Metabolic Disorder; Liver Failure, Chronic
MeSH Terms: conditions — Metabolic Diseases; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy and Cirrhosis (Other): Ammonia infusion with and without ammonia targeting
  Interventions: Other: Ammonia infusion

INTERVENTIONS:
Other: Ammonia infusion — Ammonia metabolism investigated in healthy individuals and patients with cirrhosis with and without ammonia lowering agent: glycerolphenylbutyrat (healthy) and Lactulose + Rifaximin (Cirrhosis)

SUMMARY:
The present study will develop a method to assess ammonia metabolism by ammonia infusion and investigate ammonia production and clearance in healthy individuals and in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria - Healthy controls:

* Alcohol < 40g/day
* BMI < 30
* Diseased or medicated

Inclusion Criteria - Patients with cirrhosis:

* Child-Pugh A or B cirrhosis
* BMI < 30

Exclusion Criteria:

* Child-Pugh score C
* Kidney failure (eGFR < 60 mL/min/1.73m2)
* Overt hepatic encephalopathy or more than one previous 1 episode of overt hepatic encephalopathy
* Acute bacterial infection
* Cancer
* Diabetes
* Ammonia-targeted treatment of hepatic encephalopathy other than lactulose (including Rifaximin and branched-chain amino acids)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clearance (L/min) and production (micromol/min) of ammonia | 2 years
  A physiological parameter

SECONDARY OUTCOMES:
Change in clearance (L/min) and production (micromol/min) of ammonia when measured while on ammonia modulating agents | 2 years
  Proof of concept

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology & Gastroenterology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No